CLINICAL TRIAL: NCT00734760
Title: Reducing Prehospital Delay in Acute Myocardial Infarction
Brief Title: An Intervention to Reduce Prehospital Delay to Treatment in Acute Coronary Syndrome
Acronym: PROMOTION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Kathleen Dracup, University of California, San Francisco
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RO! NR05323; NIH RO! NR05323
Record Dates: First submitted 2008-08-12; First posted 2008-08-14 (Estimated); Last update posted 2008-08-14 (Estimated); Status verified 2008-08

CONDITIONS: Acute Coronary Syndrome
Keywords: patient education; acute coronary syndrome; prehospital delay to treatment
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): a tailored, face-to-face education and counseling intervention with a nurse lasting approximately 45 minutes, followed by a telephonic reinforcement in 30 days
  Interventions: Behavioral: education
- B (No Intervention): care-as-usual with data collection at the same time points as the experimental group

INTERVENTIONS:
Behavioral: education — face-to-face education and counseling intervention
  Other Names: none applicable
  Arms: A

SUMMARY:
This study was conducted to test whether a focused education and counseling intervention delivered by a nurse will decrease time of delay in seeking treatment for the signs and symptoms of acute coronary syndrome (i.e., heart attack) in patients already identified as having ischemic heart disease.

DETAILED DESCRIPTION:
Delay to treatment from the onset acute coronary syndrome (ACS)continues to be a significant cause of morbidity and mortality. This study was conducted to evaluate a tailored education and counseling program designed for individuals at high risk for a future event. Study Hypothesis: The central hypothesis of this study was that a focused education and counseling intervention delivered by a nurse will decrease time of delay in seeking treatment for the signs and symptoms of AMI in patients already identified as having ischemic heart disease. Patients were randomized to receive a nurse-administered education and counseling intervention designed to promote early presentation for medical treatment in the face of cardiac symptoms or to usual instructions by their healthcare provider. Primary & Secondary Endpoints: The primary endpoint of this trial was prehospital delay time, i.e., time from onset of symptoms to arrival at the hospital. The secondary endpoints were: use of the emergency medical system; use of aspirin; healthcare resource utilization; and knowledge, attitudes and beliefs about heart disease.

ELIGIBILITY:
Inclusion Criteria:

* a diagnosis of ischemic heart disease, confirmed by their physician or medical record
* lived independently (i.e., not in an institutional setting).

Exclusion Criteria:

* complicating serious co-morbidity such as a psychiatric illness or untreated malignancy
* neurological disorder with impaired cognition
* inability to read or understand English.
* major uncorrected hearing loss

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3522 (Actual)
Dates: Start 2001-02; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
time from ACS symptom onset to admission to emergency department | two years

SECONDARY OUTCOMES:
pre-hospital aspirin use | two years
emergency medical system use | two years
resource utilization | two years

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen A Dracup, DNSc, Principal Investigator — University of California, San Francisco

REFERENCES:
- [Background] Dracup K, McKinley S, Doering LV, Riegel B, Meischke H, Moser DK, Pelter M, Carlson B, Aitken L, Marshall A, Cross R, Paul SM. Acute coronary syndrome: what do patients know? Arch Intern Med. 2008 May 26;168(10):1049-54. doi: 10.1001/archinte.168.10.1049. PMID 18504332
- [Background] Aitken LM, Pelter MM, Carlson B, Marshall AP, Cross R, McKinley S, Dracup K. Effective strategies for implementing a multicenter international clinical trial. J Nurs Scholarsh. 2008;40(2):101-8. doi: 10.1111/j.1547-5069.2008.00213.x. PMID 18507563
- [Background] Riegel B, McKinley S, Moser DK, Meischke H, Doering L, Dracup K. Psychometric evaluation of the Acute Coronary Syndrome (ACS) Response Index. Res Nurs Health. 2007 Dec;30(6):584-94. doi: 10.1002/nur.20213. PMID 18022812
- [Background] Dracup K, McKinley S, Riegel B, Mieschke H, Doering LV, Moser DK. A nursing intervention to reduce prehospital delay in acute coronary syndrome: a randomized clinical trial. J Cardiovasc Nurs. 2006 May-Jun;21(3):186-93. doi: 10.1097/00005082-200605000-00006. PMID 16699358
- [Derived] Dracup K, McKinley S, Riegel B, Moser DK, Meischke H, Doering LV, Davidson P, Paul SM, Baker H, Pelter M. A randomized clinical trial to reduce patient prehospital delay to treatment in acute coronary syndrome. Circ Cardiovasc Qual Outcomes. 2009 Nov;2(6):524-32. doi: 10.1161/CIRCOUTCOMES.109.852608. Epub 2009 Oct 6. PMID 20031889